CLINICAL TRIAL: NCT06960356
Title: Development of Follow-up Nursing Consultations for Children at Risk of Post-resuscitation Syndrome
Acronym: SURVIPED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC24.0249; 2024-A01670-47 (Other: RCB)
Record Dates: First submitted 2025-03-13; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-01

CONDITIONS: Stress Disorder, Post Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- screening for post-resuscitation syndrome (Experimental)
  Interventions: Other: detect post-traumatic stress disorder

INTERVENTIONS:
Other: detect post-traumatic stress disorder — recommendation for follow-up by a professional specializing in child development and/or a complementary medical consultation

SUMMARY:
The investigator hypothesize that, during an IPDE consultation 3 months after discharge from critical care, the investigator will identify PTSD in approximately one-third of children, and show an association between this syndrome and quality of life in children admitted to pediatric intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 1 and 17.5 years at inclusion
* Having stayed in a paediatric intensive care unit in one of the 2 participating centers: Lyon or Grenoble
* Requiring mechanical ventilation (invasive or non-invasive) for more than 24 hours

Exclusion Criteria:

* Patients already under the care of a psychologist or psychiatrist
* patients who died during their stay in intensive care
* Patients who died between discharge and 3 months
* Patients suspected of abuse
* Patient and/or parent refusal to participate
* No social security affiliation
* Patients / parents who do not speak French

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
post-traumatic stress disorder | 3 months
  Prevalence of post-traumatic stress disorder (PTSD) as defined by a standardized assessment of PTSD using the Children's Revised Impact of Event Scale (CRIES-13) scale for children over 7 years of age.
  Range from 0 to 80. Higher scores indicate greater post-traumatic stress

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory TM (PEDSQL scale) | 3 months
  assessing Pediatric Quality of Life Inventory TM (PESQL scale) at 3 months in patients admitted to pediatric critical care. Range from 0 to 230.
  Higher scores indicate better health related quality of life.
correlation between the PTSD score and the child's quality of life | 3 months
  correlation between the post-traumatic stress disorder score (Using Children's Revised Impact of Event Scale - range from 0 to 65 - the higher the score, the greater the impact of the event on the child) and the child's quality of life ( Using Pediatric Quality of Life Inventory TM scale - range from 0 to 230 - higher scores indicate better health-related quality of life)
Measurement of the association between the characteristics of children and their stay in critical care, and the presence of PTSD | 3 months
  Search for factors associated with the onset of PTSD. Measurement of the association between the characteristics of children and their stay in critical care, and the presence of PTSD (using the Children's Revised Impact of event Scale - Range from 0to 65 - the higher the score, the greater the impact of the event on the child)
number of children with significant somatic symptoms | 3 months
  Estimate the proportion of children presenting significant and disabling somatic symptoms in their lives, requiring referral to the appropriate healthcare professionals.
Screening parents for PTSD | 3 months
  Screening parents for PTSD using the POst-Traumatic stress disorder checklist version DSM-5 (PCL 5). range from 0 to 80 - the higher the score, the greater the post-traumatic stress
factors associated with the occurrence of PTSD in parents | 3 months
  Measurement of the association between the characteristics of the children and their stay in critical care, and the presence of PTSD in the parents with Post-Traumatic stress disorder checklist version DSM-5 (PCL 5). range from 0 to 80 - the higher the score, the greater the post-traumatic stress
Evaluate the feasibility of having the follow-up critical care consultation carried out by a nursery nurse | 3 months
  time devoted to organising and carrying out consultations and referrals, number and proportion of parents who do not attend consultations (parental involvement)